CLINICAL TRIAL: NCT01720862
Title: Migraine and Body Composition
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Drs Barbara Peterlin, Director of Headache Research, Johns Hopkins Bayview, Johns Hopkins University
Other Study IDs: NA_00051683
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Migraine With and Without Aura; Chronic Migraine; Healthy Controls
Keywords: migraine; episodic migraine; chronic migraine; obesity; non-obese
MeSH Terms: conditions — Migraine Disorders; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Episodic migraineurs: Those with migraines >2 and < 12 times per month.
- Chronic migraineurs: Those with migraines greater than 14 days per month.
- Controls: Those without headaches other than occasional hangover, cold, flu headaches.

SUMMARY:
This research is being done to look at the association between migraine and obesity.

DETAILED DESCRIPTION:
Research into the role of inflammatory markers and other obesity related proteins and chemicals may help us understand migraine and lead to new treatment.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women (18-55 years)
* Normal weight (BMI = 18.5 - 24.9) or obese (BMI ≥ 30)
* Diagnosis of episodic or chronic migraine or pain free control

Exclusion Criteria:

* Evidence of pain disorder other than migraine (e.g. irritable bowel syndrome)
* Chronic conditions known to alter risk or pattern of migraine (e.g. hypothyroidism)
* Illnesses that may affect adipokine levels (e.g. diabetes)
* Clinically relevant abnormal glucose/cholesterol levels
* Pregnant women
* Potential participants who are unable to undergo MRI based on standard screening questionnaire (those with brain aneurysm or surgical clips, certain types of artificial heart valves, heart defibrillator or pacemaker, cochlear implants, eye implants, blood vessel coil, recently placed artificial joints, certain types of vascular stents, history of bullets, pellets, BBs, history of any implanted metal or device or who have worked with sheet metal in the past)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Premenopausal Caucasian women ages 18-55 years with or without migraine.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
association between migraine and obesity - evaluate serum adipokine levels | 5 years
  The first aim of the proposed research is to evaluate serum adipokine levels in a clinical cohort of obese and non-obese episodic and chronic migraineurs and examine their utility as markers of the presence or absence of migraine and their relationship to headache frequency.

SECONDARY OUTCOMES:
association between migraine and obesity -evaluate subcutaneous adipose tissue (SAT) and its ratio to visceral adipose tissue (VAT) | five years
  The second aim of the proposed research is to evaluate subcutaneous adipose tissue (SAT) and its ratio to visceral adipose tissue (VAT),in the same clinical cohort of migraineurs to determine if regional adipose tissue differences exist between: (1) episodic migraineurs, (2) chronic migraineurs and (3) controls, thus contributing to the migraine-obesity relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara L Peterlin, DO, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Bayview Headache Center, Baltimore, Maryland, United States